CLINICAL TRIAL: NCT00762736
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Proof-of-Concept Study of the Efficacy, Safety, and Tolerability of Pioglitazone HCl (ACTOS™) in Combination With TAK-536 in Subjects With Type II Diabetes
Brief Title: Efficacy and Safety of Pioglitazone and Azilsartan in Treating Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-OPI-525; U1111-1115-8992 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Pioglitazone 15 mg QD + Azilsartan 5 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and azilsartan
- Pioglitazone 15 mg QD + Azilsartan 40 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and azilsartan
- Pioglitazone 15 mg QD (Active Comparator)
  Interventions: Drug: Pioglitazone
- Pioglitazone 45 mg QD + Azilsartan 5 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and azilsartan
- Pioglitazone 45 mg QD + Azilsartan 40 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and azilsartan
- Pioglitazone 45 mg QD (Active Comparator)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone and azilsartan — Pioglitazone 15 mg, tablets, orally, once daily and azilsartan 5 mg, tablets, orally, once daily for up to 24 weeks.
  Other Names: ACTOS®; AD4833; TAK-536
  Arms: Pioglitazone 15 mg QD + Azilsartan 5 mg QD
Drug: Pioglitazone and azilsartan — Pioglitazone 15 mg, tablets, orally, once daily and azilsartan 40 mg, tablets, orally, once daily for up to 24 weeks.
  Other Names: ACTOS®; AD4833; TAK-536
  Arms: Pioglitazone 15 mg QD + Azilsartan 40 mg QD
Drug: Pioglitazone — Pioglitazone 15 mg, tablets, orally, once daily and azilsartan placebo-matching tablets, orally, once daily for up to 24 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone 15 mg QD
Drug: Pioglitazone and azilsartan — Pioglitazone 45 mg, tablets, orally, once daily and azilsartan 5 mg, tablets, orally, once daily for up to 24 weeks.
  Other Names: ACTOS®; AD4833; TAK-536
  Arms: Pioglitazone 45 mg QD + Azilsartan 5 mg QD
Drug: Pioglitazone and azilsartan — Pioglitazone 45 mg, tablets, orally, once daily and azilsartan 40 mg, tablets, orally, once daily for up to 24 weeks.
  Other Names: ACTOS®; AD4833; TAK-536
  Arms: Pioglitazone 45 mg QD + Azilsartan 40 mg QD
Drug: Pioglitazone — Pioglitazone 45 mg, tablets, orally, once daily and azilsartan placebo-matching tablets, orally, once daily for up to 24 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone 45 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy of pioglitazone, once daily (QD), combined with azilsartan in the treatment of subjects with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Diabetes is a chronic disease with multiple metabolic defects that result in hyperglycemia arising from inadequate insulin activity. Type 2 diabetes has a genetic predisposition, but lifestyle, body constitution and age play important roles in determining its time of onset and severity. Type 2 diabetes is usually the result of a progression from reduced sensitivity of hepatic and peripheral-tissue cells to circulating insulin (i.e., insulin resistance) to a progressive inability of the body to produce adequate insulin to overcome insulin resistance (i.e., insulin deficiency due to beta cell insufficiency) resulting in impaired glucose tolerance and ultimately overt diabetes. In the United States, an estimated 15.7 million people have diabetes, with type 2 diabetes occurring in approximately 90-95% of cases.

Therapeutic agents have been developed to address each of the major functional metabolic defects associated with type 2 diabetes: decreased beta-cell function, elevated hepatic glucose output, and insulin resistance. The oral therapeutic agents used in the treatment of type 2 diabetes can be separated into the following four categories based on their mechanisms of action: insulin secretagogues, inhibitors of hepatic glucose output, inhibitors of complex carbohydrate breakdown in the intestine and insulin sensitizers.

Thiazolidinediones reduce insulin resistance by enhancing insulin sensitivity in muscle cells, adipose tissue, and hepatic cells (inhibiting hepatic gluconeogenesis) with no direct impact on insulin secretion. Thus thiazolidinediones improve glycemic control and result in reduced levels of circulating insulin. Peroxisome proliferator-activated receptors are found in tissues important for insulin action, such as adipose tissue, skeletal muscle, and the liver. The greatest concentration of peroxisome proliferator-activated receptors -gamma receptors is in adipose tissue. Pioglitazone HCl (ACTOS®) is a thiazolidinedione developed by Takeda Chemical Industries, Ltd.

Research suggests that Angiotensin II receptor blockers are involved in endothelial and cardiovascular function, and in insulin sensitization and obesity. TAK-536 (azilsartan) is an angiotensin II receptor antagonist with affinity for and selective antagonistic activity at the angiotensin II type 1 receptor.

This study was designed to evaluate the efficacy, safety, and tolerability of pioglitazone in combination with azilsartan in subjects with type 2 diabetes.

Study participation is anticipated to be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Had type 2 diabetes, with a hemoglobin value of greater than or equal to 8.0% or less than 10.0% at Screening.
* Females of childbearing potential who were sexually active agreed to use adequate contraception, and were neither pregnant nor lactating from Screening throughout the duration of the study.
* Received antihypertensive therapy and must have been on a stable dose for a minimum of 8 weeks prior to Screening.
* Had clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory unless the results were deemed not clinically significant for inclusion into this study by the investigator or sponsor.
* Had been on stable diet and exercise program and oral anti-glycemic therapy including sulfonylurea or metformin for 8 weeks prior to Screening.

Exclusion Criteria:

* Had a hemoglobin value less than 8.0% or greater than 10.0% at Screening.
* Was taking an angiotensin II receptor blocker.
* Had uncontrolled hypertension defined as systolic blood pressure greater than 160 mm Hg and diastolic blood pressure greater than 100 mm Hg. - Had a systolic blood pressure less than or equal to 110 mm Hg and/or diastolic blood pressure less than or equal to 60 mm Hg.
* Was taking or was expected to take the following medications:

  * antidiabetic agents (other than sulfonylurea or metformin)
  * tricyclic antidepressants
  * monoamine oxidase inhibitors
  * phenothiazines
  * diet medications
  * amphetamines or their derivatives
  * lithium
  * common cold medications with chronic use
  * nonsteroidal anti-inflammatory drugs with chronic use (including aspirin greater than 325 mg/day or cyclooxygenase 2 inhibitors).
* Had unstable angina or heart failure of any etiology with functional class New York Heart Association III or IV.
* Had a history of myocardial infarction.
* Had clinically significant cardiac conduction defects (eg, second or third degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation or flutter).
* Had secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
* Had a history of collagen vascular disorder (eg, systemic lupus erythematosus, scleroderma) within the last 5 years.
* Had a body mass index greater than 39 kg/m2.
* Had significant, moderate-to-severe renal dysfunction (creatinine greater than 2.4 mg/dL). If receiving metformin, a creatinine greater than 1.5 mg/dL for male subjects or greater than 1.4 mg/dL for female subjects led to exclusion.
* Had a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Had a previous history of cancer, other than basal cell carcinoma, that had not been in remission for at least 5 years prior to the first dose of study drug.
* Had type 2 diabetes with clinically important retinopathy or peripheral or autonomic neuropathy.
* Had an alanine aminotransferase or aspartate aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
* Was participating in another investigational study or had participated in an investigational study within 30 days prior to randomization.
* Had any other serious disease or condition at Screening (or randomization) that might have compromised subject safety, affected life expectancy, or made it difficult to successfully manage and follow the subject according to the protocol.
* Was hypersensitive to angiotensin II receptor blockers.
* Was hypersensitive to thiazolidinediones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2004-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in glycosylated hemoglobin. | Week 24 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in glycosylated hemoglobin. | Weeks 12, 16, 20, and 24 or Final Visit
Change from Baseline in fasting plasma glucose. | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in total cholesterol. | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in high-density lipoprotein. | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in low-density lipoprotein. | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in triglycerides. | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in body weight. | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in systolic and diastolic blood pressure. | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in incidence of edema (peripheral). | Weeks 2, 4, 6, 8. 12, 16, 20, and 24 or Final Visit
Change from Baseline in microalbuminuria excretion. | Week 24 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein. | Weeks 12 and 24 or Final Visit
Change from Baseline in matrix metalloproteinase-9. | Weeks 12 and 24 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (78):
- United States (64):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Sierra Vista, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Burbank, California
  - Escondido, California
  - Irvine, California
  - La Jolla, California
  - National City, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - Spring Valley, California
  - Coral Gables, Florida
  - DeLand, Florida
  - Hollywood, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Opa-locka, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Warner Robins, Georgia
  - Honolulu, Hawaii
  - Lihue, Hawaii
  - Chicago, Illinois
  - Dyersburg, Indiana
  - Overland Park, Kansas
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Salisbury, Massachusetts
  - Cadillac, Michigan
  - Detroit, Michigan
  - Livonia, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - North Las Vegas, Nevada
  - Berlin, New Jersey
  - Blackwood, New Jersey
  - Trenton, New Jersey
  - Albany, New York
  - Kingston, New York
  - Charlotte, North Carolina
  - Marion, Ohio
  - Clinton, Oklahoma
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scotland, Pennsylvania
  - Woonsocket, Rhode Island
  - Greer, South Carolina
  - Arlington, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Midland, Texas
  - North Richard Hills, Texas
  - San Antonio, Texas
  - Renton, Washington
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - Rosario-Santa Fe
  - Santa Fe
  - Ushuaia - Tierre Del Fuego
- Santiago, Chile
- Mexico (6):
  - Aguascalientes
  - Cuernavaca
  - Durango
  - Guadalajara
  - Mexico City
  - Puebla City
- Peru (2):
  - Ica
  - Lima

REFERENCES:
- See also: Actos Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI